CLINICAL TRIAL: NCT06054360
Title: Predictive Value of Right Atrial Strain in Postoperative Atrial Fibrillation in Patients Undergoing Cardiac Surgery
Acronym: ODFAPO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2023_843_0048
Record Dates: First submitted 2023-09-19; First posted 2023-09-26 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Postoperative Atrial Fibrillation; Strains
Keywords: coronary bypass grafting; postoperative atrial fibrillation; strain; left atrial; right atrial
MeSH Terms: conditions — Sprains and Strains

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The incidence of postoperative atrial fibrillation (POAF) after cardiac surgery is around 30%. POAF increases the risk of developing permanent atrial fibrillation and raises the risk of cardiac decompensation, stroke, acute myocardial infarction, and death. While the role of the left atrium (LAF) in the pathophysiology of POAF is now well-established, the part of the right atrium (RA) remains poorly understood. Recent studies suggest a correlation between RA function and POAF.

RA function can be assessed by transthoracic echocardiography (TTE) with dedicated software for measuring the RA strain (RAS). RA function is thus divided into three phases: reservoir (RASr), conduit, and contraction. Numerous studies have demonstrated that a significant alteration in RAS predicts POAF in various clinical contexts. Therefore, it is essential to investigate whether alterations in RA function assessed by 2D-STE (RAS) are associated with an increased occurrence of FAPO after cardiac surgery.

It is essential to investigate whether alterations in RA function assessed by 2D-STE (RAS) are associated with an increased occurrence of FAPO after cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (>18 years old)
* The patient was hospitalized at the Amiens University Hospital for scheduled aortocoronary bypass grafting under cardiopulmonary bypass.
* Echocardiographic image quality enabling the measurement of RAS parameters
* Patient affiliation to a social security scheme
* Patient/proxy information and collection of their non-opposition.

Exclusion Criteria:

* Patients participating in an interventional study may modify the incidence of POAF.
* History of atrial fibrillation or flutter.
* Valvular and ascending aorta cardiac surgery
* Urgent cardiac surgery.
* Presence of tricuspid insufficiency greater than grade 2.
* Left ventricular ejection fraction lower than 50%.
* Patient receiving circulatory mechanical assistance before surgery.
* Dependency on ventricular and atrial pacing by an internal or external cardiac pacemaker during the echocardiographic examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This prospective, single-center study was conducted at the Amiens University Hospital. As an additional procedure to the patient's management, it includes the systematic performance of a TTE the day before the surgery, with the acquisition of specific views to measure RAS. After enrollment, the principal investigator will perform a TTE to measure RASr on particular views. TTE will be performed in a supine position at the patient's bedside by a trained medical operator, following a standardized protocol. After surgery, the patient will be monitored by a 5-lead ECG to diagnose POAF. The maximum duration of POAF monitoring will be seven days in the intensive care unit.
Sampling Method: Non-Probability Sample
Enrollment: 334 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Correlation of RASr parameter variation with POAF incidence | 30 months
  Correlation of RASr parameter variation with POAF incidence in patients undergoing postoperative cardiac surgery

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, France

IPD SHARING:
Plan to Share IPD: No